CLINICAL TRIAL: NCT01390688
Title: Brain-derived Neurotrophic Factor: A Link to Obesity, Insulin Resistance and Cognitive Dysfunktion?
Brief Title: Brain-derived Neurotrophic Factor and Cogntive Function
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Maria Pedersen/ MD, Centre of Inflammation and Metabolism
Other Study IDs: H-4-2011-031
Record Dates: First submitted 2011-07-05; First posted 2011-07-11 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2009-06

CONDITIONS: Cognitive Dysfunction; Glucose Metabolism; Low-grade Inflammation; Bodycomposition
Keywords: Brain-derived Neurotrophic factor; Low-grade inflammation; Cognitive dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, Serum, DNA, Muscle tissue and fat tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Type 2 Diabetes: 80 individuals with type 2 Diabetes, confirmed by an OGTT, age 40-65 years, BMI > 18.5 kg/m2 fatsing plasma glucose < 12 mmol/l
- Impaired glucose tolerance: 40 individuals with impaired glucose tolerance. age 40 -65 years, BMI > 18. 5 kg/m2
- Normal glucose tolerance: 80 Individuals without type 2 diabetes Age 40-65 years, BMI >18.5 kg/m2.

SUMMARY:
Individuals with type 2 diabetes have an increased risk of developing cognitive dysfunction followed by dementia in late life. Obesity, physical inactivity and "systemic low-grade inflammation" are strong risk factors and play a crucial role in this network of diseases.

Brain-derived Neurotrophic factor (BDNF) is produced in brain as well as several tissues outside brain eg muscle cells. Low BDNF are associated with cognitive dysfuction, obesity and type 2 diabetes.

The investigators include 200 individuals divided into three groups: 80 individuals with type 2 diabetes, 80 age and BMI-matched controls and 40 individuals with impaired glucose tolerance.

The project will test the hypothesis, that low systemic BDNF are associated with accumulation of abdominal fat, cognitive dysfunction and insulin resistence with different effect in men and women.

DETAILED DESCRIPTION:
Methods:

200 individuals in age 40-65 years are recruited and categorized into 3 groups: 1. Type 2 Diabetes, 2. Impaired glucose Tolerance and 3. Normal Glucose Tolerance. Groups are supposed to be age and BMI-matched.

Measurements of systemic BDNF, cogntive function (memory, attention and langue), fitness, bodycomposition, glucose metabolism and systemic inflammation are done.

Multiple regression analysis are perfomed to explain variablity in cognitive function, with age, visceral fat and BDNF as explanotory varibales.

ELIGIBILITY:
Inclusion Criteria:

* 40-65 years of age

Exclusion Criteria:

* Chronic inflammatory diseases or infectious diseaases within 3 month prior to visit
* Fasting glucose > 12 mmol/l
* Hypertension: systolic >180 mmHg and Diastolic >110 mmHg
* Intake of more than 2 oral antidiabetic drugs or any TZD drung within 3 months before recruitment

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from newspapers.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Systemic Brain derived neurotrophic factor | Baseline
  Circulating Brain derived neurotropic factor will be analyzed in plasma and serum in middelaged volunteers. Levels will be related to on one hand metabolic parameteres such as insulin sensitivity and glucose tolerance and on the other hand to cognitive functions measured by a cognitive test battery.

SECONDARY OUTCOMES:
Cognitive function and bodycompisition | Baseline
  Results from cogntive measurements will by multiple regression analysis be related to bodycomposition (Intraabdominal fat, total bodyfat, waist) and fitness (single stage max-test).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Inflammation and Metabolism, Copenhagen, Denmark